CLINICAL TRIAL: NCT01635608
Title: Absorption of Paracetamol, Talinolol and Amoxicillin After Oral Administration Using Non-caloric and Caloric Water
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MRI-probe drugs; 2011-000228-13 (EudraCT Number)
Record Dates: First submitted 2012-07-04; First posted 2012-07-09 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Gastrointestinal Motility Disorder
Keywords: Pharmacokinetics; Talinolol; Amoxicillin; Acetaminophen; Magnetic Resonance Imaging
MeSH Terms: interventions — Acetaminophen; talinolol; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- non-caloric water (Active Comparator): 500 mg paracetamol, 50 mg talinolol and 500 mg amoxicillin dissolved in 240 ml non-caloric water immediately before administration after overnight fasting
  Interventions: Drug: Acetaminophen; Drug: Talinolol; Drug: Amoxicillin; Other: non-caloric water
- caloric water (Active Comparator): 500 mg paracetamol, 50 mg talinolol and 500 mg amoxicillin dissolved in 240 ml caloric water immediately before oral administration after overnight fasting
  Interventions: Drug: Acetaminophen; Drug: Talinolol; Drug: Amoxicillin; Other: caloric water

INTERVENTIONS:
Drug: Acetaminophen — administration of 500 mg paracetamol
Drug: Talinolol — administration of 50 mg talinolol
Drug: Amoxicillin — administration of 500 mg amoxicillin
Other: non-caloric water — administration of 240 ml water
  Arms: non-caloric water
Other: caloric water — administration of 240 ml caloric water (containing 25.5 g sucrose)
  Arms: caloric water

SUMMARY:
To visualize the localization and to measure the volume of water in the small intestine by T2-weighted MRI imaging after oral administration of 240 ml water (non-caloric water) and after administration of 240 ml water containing 25.5 g sucrose (105 kcal, caloric water).

To measure pharmacokinetics of the probe-drugs paracetamol, talinolol and amoxicillin after oral administration dissolved in 240 ml non-caloric and in 240 ml caloric water.

DETAILED DESCRIPTION:
After swallowing, a drug first is deposited in the stomach together with the co-swallowed water. However, the stomach is not the major place of drug absorption. Therefore, the kinetics of gastric emptying plays a crucial role for the absorption process. In case of dissolved or finely suspended drug particles, gastric emptying of the drugs occurs together with gastric contents. The emptied liquid enters the small intestine where it is absorbed. Under fasting conditions, the emptied phase consists of the water that was co-swallowed with the drug (in clinical studies typically 240 ml) together with a small volume of gastric juice. Under fed conditions, the emptied liquid phase is a caloric suspension. It is known that both the gastric emptying and the intestinal absorption of pure water are rapid leading usually to rapid absorption of water soluble drugs that are taken under fasting conditions. In the contrary, delayed absorption under postprandial conditions is typically related to delayed gastric emptying. However, velocity and extent of intestinal filling and the absorption rate of the liquid phase from gut lumen are unknown.

Therefore, it is the primary objective of the study to determine the gastric emptying kinetics of 240 ml water (non-caloric water) and of 240 ml water containing 25.5 g sucrose (105 kcal, caloric water), the respective intestinal filling and the absorption rate of the intestinal liquid using water sensitive magnetic resonance imaging (MRI).

To evaluate the functional meaning of gastric emptying, intestinal filling and water uptake for oral drug absorption which are swallowed with non-caloric and caloric water, pharmacokinetics of paracetamol, talinolol and amoxicillin will be studied after administration with 240 ml non-caloric and 240 ml caloric water, respectively.

Paracetamol (acetaminophen) was chosen, because it is rapidly and completely absorbed from all parts of the gut. The time of its appearance in blood is expected to be a surrogate for the rate of gastric emptying. It is hypothesized that caloric content of the water for administration does not influence the extent of paracetamol absorption.

Talinolol represents a well established probe drug for the intestinal efflux transport protein ABCB1. Because expression of ABCB1 increases along the small intestine (duodenum<jejunum<ileum), we hypothesize, that administration of talinolol with caloric water leads to lower bioavailability and increase of the fecal excretion of the drug.

Amoxicillin acts as a probe drug for intestinal drug uptake via the dipeptide transporter PEPT1 which is predominately expressed in proximal parts of the small intestine ((duodenum>jejunum>ileum). Because of this region-specific expression, we hypothesize, that administration of amoxicillin with caloric water is associated with lower bioavailability.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 - 45 years
* sex: male and female
* ethnic origin: white
* body weight between 19 and 27 kg/m²
* good health as evidenced by the results of the clinical examination, ECG, and the laboratory check-up, which are judged by the clinical investigator not to differ in a clinical relevant way from the normal state
* written informed consent

Exclusion Criteria:

* weight less than 45 kg
* claustrophobia
* cardiac pacemakers, metallic implants or metal-containing tatoos
* known allergic reactions to the active ingredients used or to constituents of the study medication
* bronchial asthma (all stages)
* existing cardiac or hematological diseases and/or pathological findings, which might interfere with the drug's safety, tolerability and/or pharmacokinetics (e.g. tachycardia)
* hepatic and renal diseases and/or pathological findings, which might interfere with pharmacokinetics and pharmacodynamics of the study medication
* gastrointestinal diseases and/or pathological findings, which might interfere with pharmacokinetics and pharmacodynamics of the study medication
* drug or alcohol dependence
* positive drug or alcohol screening
* smokers of 10 or more cigarettes per day
* positive results in HIV, HBV and HCV screenings
* subjects who are on a diet which could affect the pharmacokinetics of the drug
* heavy tea or coffee drinkers (more than 1L per day)
* lactation and pregnancy test positive or not performed
* subjects suspected or known not to follow instructions
* subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to as a result of their participation in the study
* subjects liable to orthostatic dysregulation, fainting, or blackouts
* participation in a clinical trial during the last 3 months prior to the start of the study
* less than 14 days after last acute disease
* less than 3 months after last blood donation
* any systemically available medication within 2 weeks prior to the intended first administration unless because of the terminal elimination half-life complete elimination from the body can be assumed for the drug and/or its primary metabolites (except oral contraceptives)
* intake of grapefruit or poppy seeds containing products within 14 days prior to administration

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-04; Primary Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Correlation between volume of water in stomach and AUC of study medication | 0 to 48 h

SECONDARY OUTCOMES:
area under the concentrations-time curve (AUC) | 0, 5, 10, 15, 20, 30, 40, 50, 60, 75, 90, 105 min and 2, 3, 4, 6, 8, 12, 24 and 48 h after drug administration
maximum concentration (Cmax) | 0, 5, 10, 15, 20, 30, 40, 50, 60, 75, 90, 105 min and 2, 3, 4, 6, 8, 12, 24 and 48 h after drug administration
volumen of water in stomach | before and 1.5, 6.5, 11.5, 16.5, 21.5, 26.5, 31.5, 36.5, 41.5, 46.5, 51.5, 56.5, 61.5, 66.5, 71.5, 76.5, 81.5, 86.5, 91.5, 96.5, 101.5, 106.5, 111.5, and 116.5 min after administration of the study medication
  Dynamic enhanced MR examination gradient-echo T2-weighted HASTE images (TR 1900 ms, TR 111 ms, flip-angle 0) will be acquired on a 1.5T MRI. A tube filled with 20 ml water will be fitted on the abdomen of the volunteers in order to have an internal reference for imaging.
volumen of water in small intestine | before and 1.5, 6.5, 11.5, 16.5, 21.5, 26.5, 31.5, 36.5, 41.5, 46.5, 51.5, 56.5, 61.5, 66.5, 71.5, 76.5, 81.5, 86.5, 91.5, 96.5, 101.5, 106.5, 111.5, and 116.5 min after administration of the study medication
  Dynamic enhanced MR examination gradient-echo T2-weighted HASTE images (TR 1900 ms, TR 111 ms, flip-angle 0) will be acquired on a 1.5T MRI. A tube filled with 20 ml water will be fitted on the abdomen of the volunteers in order to have an internal reference for imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Ernst-Moritz-Arndt-University Greifswald, Greifswald, Meckleburg-Vorpommern, Germany